CLINICAL TRIAL: NCT04522765
Title: Diurnal Blood Pressure and Arterial Stiffness Patterns in Those at Increased Risk of Cardiovascular Disease
Brief Title: Diurnal BP Patterns in Those at Increased Risk of CVD
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC19178
Record Dates: First submitted 2020-08-14; First posted 2020-08-21 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Risk Factor; Blood Pressure; Arterial Stiffness; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Blood Pressure; Vascular Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples will be obtained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Health: Healthy individuals with no known medical condition and taking no regular medication
  Interventions: Diagnostic Test: Assessment of 24 hour blood pressure and arterial stiffness
- Acute kidney injury: Individuals with acute kidney injury as defined by KDIGO criteria
  Interventions: Diagnostic Test: Assessment of 24 hour blood pressure and arterial stiffness
- Chronic kidney disease: Individuals with chronic kidney disease as defined by KDIGO criteria
  Interventions: Diagnostic Test: Assessment of 24 hour blood pressure and arterial stiffness
- Small vessel vasculitis: Individuals with active small vessel vasculitis an diagnosed by a specialist physician
  Interventions: Diagnostic Test: Assessment of 24 hour blood pressure and arterial stiffness
- Kidney transplant recipient: Individuals who have received a kidney transplant
  Interventions: Diagnostic Test: Assessment of 24 hour blood pressure and arterial stiffness
- Kidney donor: Individuals who have donated a kidney for transplantation
  Interventions: Diagnostic Test: Assessment of 24 hour blood pressure and arterial stiffness

INTERVENTIONS:
Diagnostic Test: Assessment of 24 hour blood pressure and arterial stiffness — Assessment of 24 hour blood pressure and arterial stiffness using Mobil-o-graph device

SUMMARY:
In health, blood pressure (BP) falls at night by >10% compared with day-time values. This natural dipping pattern is important as without it there is an increased risk of cardiovascular disease (CVD). Recent evidence suggests that chronotherapy (taking anti-hypertensive medication at bedtime instead of in the morning) may enhance nocturnal BP dipping and reduce the risk of CVD events. There is therefore an urgent need to characterise diurnal BP patterns in patients who may be at risk of reduced nocturnal dipping in order to maximise protective therapy in all those who would benefit. Similarly, it has previously been demonstrated that increased arterial stiffness is associated with increased CVD risk, however little is known about whether loss of diurnal variations in arterial stiffness confer addition risk. Kidney disease is independently associated with increased CVD events, but the exact makeup of this risk is not clear. Within this heterogenous cohort several very distinct groups exist including those with acute kidney injury (AKI), chronic kidney disease (CKD), inflammatory conditions like small vessel vasculitis (SVV), and those who have either donated or received a kidney transplant. Diurnal BP and arterial stiffness patterns within these patient groups are not well characterised. The investigators will recruit patients at increased risk of CVD from the Royal Infirmary of Edinburgh Renal and Vasculitis Clinics. Participants will undergo 24-hour ambulatory BP and arterial stiffness measurement in conjunction with day- and night-time blood and urine sampling on two separate occasions. This study aims to characterise diurnal patterns of BP and arterial stiffness in patients at increased risk of CVD and compare findings with healthy controls. In doing so, the investigators aim to allow more targeted CVD risk reduction strategies and improve long-term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to take part in the study if they attend NHS Lothian inpatient or outpatient services and can be classified as being at increased risk of CVD. This will include, but is not limited to, the following subgroups:

  1. CKD as defined by the Kidney Disease Outcome Quality Initiative (K/DOQI) classification
  2. AKI as defined by the Kidney Disease Improving Global Outcomes (KDIGO) classification
  3. Small vessel vasculitis
  4. Kidney transplant recipient
  5. Kidney donor We will also recruit a healthy control group from the community.

Exclusion Criteria:

1. Age <18 years and >90 years
2. Lack of ability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Nocturnal BP dip | 24 hours
  Percentage change between mean day-time and mean night-time blood pressure
Nocturnal arterial stiffness dip | 24 hours
  Percentage change between mean day-time and mean night-time arterial stiffness

SECONDARY OUTCOMES:
Change in urine ET-1 concentration when measured in the morning (06:00 - 12:00) and in the evening (18:00-00:00) | Morning (06:00-12:00) and evening (18:00-00:00)
  Measurement of urine ET-1 concentration in the morning (06:00 - 12:00) and in the evening (18:00-00:00)
Change in plasma ET-1 concentration when measured in the morning (06:00 - 12:00) and in the evening (18:00-00:00) | Morning (06:00-12:00) and evening (18:00-00:00)
  Measurement of plasma ET-1 concentration in the morning (06:00 - 12:00) and in the evening (18:00-00:00)

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, MBChB PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD